CLINICAL TRIAL: NCT01337908
Title: A Survey of Vulnerability Factors, Current Stress and Depression Risk in Spinal Cord Injury
Brief Title: A Study of Mood and Stress After Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Wayne State University (Other); Santa Clara Valley Health & Hospital System (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Claire Z. Kalpakjian, Assistant Professor, University of Michigan
Other Study IDs: H133G070020
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Spinal Cord Injury; Depression
Keywords: depression; quality of life; disability
MeSH Terms: conditions — Spinal Cord Injuries; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Saliva samples collected with Oragene kit.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a study of factors, such as pain, family support, psychological history and alcohol/substance use, that may influence whether a person experiences depression after their spinal cord injury.

DETAILED DESCRIPTION:
The objective of this study is to examine the degree to which vulnerability factors are mediated by stress to increase risk for depression after SCI in a sample of adults who sustained their injuries after the age of 18 years. Participants will complete a written survey (about pain, daily activities, social support and life experiences) and a telephone interview that will provide information about these factors.

ELIGIBILITY:
Inclusion Criteria:

* Have a spinal cord injury
* Were age 16 years or older when injured
* Sudden onset of symptoms

Exclusion Criteria:

* Under 19 years old
* Less than 1 year post-injury
* had a non-traumatic injury

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women with a traumatic spinal cord injury who are 18 years of age and older
Sampling Method: Probability Sample
Enrollment: 377 (Actual)
Dates: Start 2009-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Santa Clara Valley Medical Center, San Jose, California
  - University of Michigan, Ann Arbor, Michigan
  - Rehabilitation Institute of Michigan, Detroit, Michigan
  - University of Washington, Seattle, Washington